CLINICAL TRIAL: NCT02703129
Title: Nutritional Intervention Fin Migraine: A 12-week Open Study
Brief Title: Nutritional Intervention in Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Antonio L Teixeira Jr, PhD, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 0311.0.203.000-11
Record Dates: First submitted 2016-02-05; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Migraine
Keywords: Migraine; Diet quality; Nutritional intervention; Severity of disease; Depressive symptoms
MeSH Terms: conditions — Migraine Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nutritional intervention (Experimental): Women with the diagnosis of migraine received individualized diet meal plan and nutritional orientations for three months according to their nutritional diagnosis
  Interventions: Other: Nutritional intervention

INTERVENTIONS:
Other: Nutritional intervention — Women with the diagnosis of migraine received individualized diet meal plan and nutritional orientations for three months according to their nutritional diagnosis

SUMMARY:
Migraine is a common medical condition. Several studies suggest that obesity and/or weight gain are risk factors for aggravating migraine course, especially increase the frequency of headache episodes. The aim of the current study was to evaluate whether nutritional intervention would be able to improve clinical parameters (as assessed by MIDAS and HIT) of patients with migraine.

DETAILED DESCRIPTION:
Women with the diagnosis of migraine according to the International Headache Society (IHS-2) criteria received individualized diet meal plan and nutritional orientation for 12 weeks according to their nutritional diagnosis. Patients were evaluated three times with an interval of 30 days between each visit. Clinical, anthropometric measurements (weight, height, waist circumference and body composition assessed by bioelectrical impedance analysis) and food evaluations were performed. Nutritional orientations were strengthened in each visit. The diet prescription did not change during intervention period. The diet quality of the patients was assessed through the Brazilian Healthy Eating Index - Revised (BHEI-R) version. Migraine severity was assessed with the Headache Impact Test (HIT) and the Migraine Disability Assessment Scale (MIDAS). Depressive symptoms were also evaluated with the Beck Depression Inventory (BDI).

ELIGIBILITY:
Inclusion Criteria:

* Women;
* Older than 18 years;
* Migraine diagnosis;
* Agree to sign the informed consent.

Exclusion Criteria:

* Patients with headaches not characterized as migraine;
* Pregnant or lactating women.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in clinical parameters of migraine patients by nutritional intervention in the last month. | 4 weeks
  Migraine impact/severity in the last month was assessed by HIT-6.
Change in clinical parameters of migraine patients by nutritional intervention in the last three month. | 12 weeks
  Migraine impact/severity in the last three month was assessed by MIDAS.

SECONDARY OUTCOMES:
Change in diet quality of migraine patients by nutritional intervention assessed with the Brazilian Healthy Eating Index - Revised (BHEI-R) | 12 weeks
  Diet quality was assessed through the Brazilian Healthy Eating Index - Revised (BHEI-R)
Change in depressive symptoms in migraine patients by nutritional intervention assessed with the Beck Depression Inventory (BDI) | 12 weeks
  Depressive symptoms were assessed by the Beck Depression Inventory (BDI)

CONTACTS AND LOCATIONS:
Overall Officials: Adaliene VM Ferreira, PhD, Study Director — Federal University of Minas Gerais; Aline Bárbara P Costa, Ms, Study Chair — Federal University of Minas Gerais; Antônio L Teixeira, PhD, Principal Investigator — Federal University of Minas Gerais; Laís B Martins, Ms, Study Chair — Federal University of Minas Gerais
Locations (1):
- Ambulatório Bias Fortes, Belo Horizonte, Minas Gerais, Brazil